CLINICAL TRIAL: NCT05521490
Title: Combating Physical Inactivity Pandemic by Promoting Physical Fitness Education and Physical Activity-Embedded Curriculum in Kindergartens
Brief Title: Combating Physical Inactivity Pandemic in Kindergartens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Baptist University (Other); Chinese University of Hong Kong (Other); Education University of Hong Kong (Other); The Hong Kong Polytechnic University (Other); Sun Yat-sen University (Other); Georgia State University (Other); Physical Fitness Association of Hong Kong, China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HK-KIDFIT
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Physical Activity; Cardiorespiratory Fitness
Keywords: Childhood Physical Inactivity; Childhood Obesity
MeSH Terms: conditions — Motor Activity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control (Other): Children allocated to the control group will continue with their usual curriculum, which includes the stipulated 30 minutes of daily physical activity.
  Interventions: Other: Usual Care Control
- Physical Activity Enhanced Curriculum (Experimental): Children allocated to the intervention group will receive enhanced physical fitness and healthy lifestyle education and a physical activity enhanced curriculum during their school year.
  Interventions: Behavioral: Physical Activity Enhanced Curriculum

INTERVENTIONS:
Other: Usual Care Control — 30 minutes of physical activity on each school day.
  Arms: Usual Care Control
Behavioral: Physical Activity Enhanced Curriculum — Additional 2.5 hours of physical activity per week in addition to the stipulated 30 minutes of daily physical activity.
  Arms: Physical Activity Enhanced Curriculum

SUMMARY:
The aim of this study is to examine the effects of a kindergarten-based, parent-involved intervention during the upper kindergarten year (K3) on physical activity and physical fitness in preschool children.

DETAILED DESCRIPTION:
This study is a two-arm cluster randomized controlled trial. Kindergartens will be randomly allocated to two groups: the usual care group and the intervention group. The usual care group will continue with their usual curriculum, which includes 30 minutes of daily physical activity stipulated by the Hong Kong SAR Government's Education Bureau. The intervention group will receive an additional 2.5 hours of physical activity per week in addition to the stipulated 30 minutes of daily physical activity. Outcome measures will be examined at baseline, 10 months (post-intervention), and 16 months (follow-up).

ELIGIBILITY:
Inclusion Criteria

1. Children aged 5-6 years (limited number of children may be between 4-5 and 6-7 years)
2. Able to communicate in Chinese
3. Able to participate in physical activity in a standard kindergarten setting

Exclusion Criteria:

1. Inherent or serious disease limiting participation in physical activity (e.g., congenital heart disease, pediatric cancer, Down syndrome).
2. Diagnosed mental illness impairing daily behavior and performance (e.g., anxiety disorder, depression, attention deficit hyperactivity disorder, psychotic disorders, autism spectrum disorder).
3. Physical disability (e.g., physical handicap, assistive device to walk).
4. Visual or hearing impairment.
5. Cognitive deficit or intellectual disability that requires special care and educational needs (e.g., handicapped children with learning difficulties).

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3300 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity | Baseline and 10 months
  Physical activity will be assessed using an actigraph device with a three-axis accelerometer.
Change in Cardiorespiratory Fitness | Baseline and 10 months
  Cardiorespiratory fitness will be assessed using the 20-meter shuttle run test.

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline and 16 months
  Physical activity will be assessed using an actigraph device with a three-axis accelerometer.
Change in Cardiorespiratory Fitness | Baseline and 16 months
  Cardiorespiratory fitness will be assessed using the 20-meter shuttle run test.
Change in Muscular Strength | Baseline, 10 months, and 16 months
  Muscular strength will be assessed using a handgrip dynamometer.
Change in Flexibility | Baseline, 10 months, and 16 months
  Flexibility will be assessed using the sit-and-reach test.
Change in Agility | Baseline, 10 months, and 16 months
  Agility will be assessed using a 4 x 10-meter shuttle run test.
Change in Balance Ability | Baseline, 10 months, and 16 months
  Balance ability will be assessed by the number of successful steps performed on a balance beam.
Change in Muscle Power | Baseline, 10 months, and 16 months
  Muscle power will be assessed using a vertical jump and a stationary long jump test.
Change in Body Mass Index | Baseline, 10 months, and 16 months
  Weight and height will be assessed using a calibrated electronic digital weighing scale and stadiometer respectively.
Change in Waist Circumference | Baseline, 10 months, and 16 months
  Waist circumference will be assessed using an inelastic measuring tape to the nearest 0.1cm.
Change in Body Fat | Baseline, 10 months, and 16 months
  Body fat will be assessed using a bioelectrical impedance-based multi-frequency segmental body composition analyzer (MC780, Tanita, Japan).
Change in Fat-Free Mass | Baseline, 10 months, and 16 months
  Fat-free mass will be assessed using a bioelectrical impedance-based multi-frequency segmental body composition analyzer (MC780, Tanita, Japan).
Change in Sedentary Behavior and Screen Time | Baseline, 10 months, and 16 months
  Sedentary behavior and screen time will be assessed using a 7-day activities logbook and accelerometer data.
Change in Treatment Self-Regulation Questionnaire Score | Baseline, 10 months, and 16 months
  Treatment Self-Regulation Questionnaire (TSRQ) will be used to assess the children's autonomous motivation and beliefs on active healthy lifestyles. The items in TSRQ will be answered on a 3-point Likert scale with a higher score corresponding to greater autonomous motivation.
Change in Theory of Planned Behavior Scale Score | Baseline, 10 months, and 16 months
  Theory of Planned Behavior Scale (TPBS) will be used to assess the children's social cognitive beliefs of health and physical activity behavior. The items in TPBS will be answered on a 3-point Likert scale with a higher score corresponding to a greater willingness to engage in the mentioned behaviors.
Change in Kiddy-KINDL | Baseline, 10 months, and 16 months
  Kiddy-KINDL will be used to assess the health-related quality of life in children.
Change in Early Development Instrument | Baseline, 10 months, and 16 months
  Early Development Instrument (EDI) will be used to assess the children's general well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Parco M Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.

REFERENCES:
- [Derived] Au WW, Leung CK, Lin SH, Yu AP, Fong DY, Wong SHS, Chan DKC, Capio CM, Yu CCW, Wong SWS, Chen YJ, Thompson WR, Siu PM. Effects of a physical activity-enhanced curriculum on increasing physical activity and improving physical fitness in preschoolers: Study protocol for a cluster randomized controlled trial (KID-FIT study). J Exerc Sci Fit. 2025 Apr;23(2):122-132. doi: 10.1016/j.jesf.2025.03.001. Epub 2025 Mar 13. PMID 40206326